CLINICAL TRIAL: NCT04588636
Title: Behavioral Therapy and Self-care vs Thermoformed Occlusal Splints in the Treatment of Masticatory Muscles Pain: a Controlled Clinical Trial.
Brief Title: Behavioral Therapy and Self-care vs Thermoformed Occlusal Splints in the Treatment of Masticatory Muscles Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Javier Salinas Aguilar, Dental surgeon, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10.17605/OSF.IO/9XTMD
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Myalgia of Mastication Muscle
Keywords: temporomandibular Joint Disorders; myalgia; occlusal splints; cognitive behavioral therapy; pain management
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia; Agnosia

STUDY DESIGN:
Intervention Model Description: To protect the blinding of the study, it was carried out by two operators: A (examiner) and B (therapist). The treatment of the subjects consisted of 5 sessions: (1) evaluation and diagnosis of recruited subjects, and taking an impression of the upper jaw by operator A; (2) teaching BST and delivery of OS by operator B; (3) first treatment control and BST booster at 2 weeks; (4) second treatment control and BST booster at 6 weeks; (5) third control of treatment and removal of OS if it corresponds to 10 weeks. All controls were performed by operator A in order to use a blind design without the knowledge of the outcome assessor. To protect this, it is explained to the subject that operator A cannot know the treatment that was delivered. Operator B delivered the treatments at random among the subjects selected by operator A after the initial examination, being himself in charge of contacting them and delivering the corresponding treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the first session, operator A explained to the study subjects the alternatives, benefits and possible complications of the treatments, but it was indicated that at the time of delivery of the treatment it would not be explained to them in which group they were assigned in order to protect blinding of treatments. Operator B was in charge of delivering the treatments randomly among the subjects selected by operator A. Finally, the controls were carried out by operator A in order to protect the blinding by not knowing the treatments of the patients at the time controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Behavioral and self-care therapy control group (Active Comparator): Subjects received verbal and written information on the etiology and prognosis of TMDs. In addition, advice on habits and behavior changes, relaxation techniques, sleep hygiene, diet modification, thermotherapy, encouragement to practice social and aerobic activities, and how to prevent risk factors and bad habits.
  Interventions: Behavioral: behavioral and self-care therapy
- Rigid occlusal splint group (Active Comparator): Subjects in this group received behavioral and self-care therapy, in combination with a rigid occlusal splint
  Interventions: Behavioral: behavioral and self-care therapy; Device: rigid occlusal splint (ROS)
- Soft occlusal splint group (Active Comparator): Subjects in this group received behavioral and self-care therapy, in combination with a soft occlusal splint
  Interventions: Behavioral: behavioral and self-care therapy; Device: soft occlusal splint (SOS)
- Non-occlusive splint group (Placebo Comparator): Subjects in this group received behavioral and self-care therapy, in combination with a non-occlusive splint
  Interventions: Behavioral: behavioral and self-care therapy; Device: non-occlusive splint (NOS)

INTERVENTIONS:
Behavioral: behavioral and self-care therapy — It is based on the premise that cognition, the process of acquiring knowledge and forming beliefs, is a primary determinant of mood and behavior. The therapy uses behavioral and self-care techniques to identify, correct and prevent behaviors or situations capable of altering the subject's state
  Other Names: BST
Device: rigid occlusal splint (ROS) — Occlusal splint formed in a vacuum from rigid individual sheets of 2 mm thick polyethylene terephthalate (Biolon, Dreve, Unna, Germany).
  Other Names: ROS
  Arms: Rigid occlusal splint group
Device: soft occlusal splint (SOS) — Occlusal splint formed in a vacuum from 3 mm thick individual soft sheets of ethyl vinyl acetate (Drufosoft, Dreve, Unna, Germany).
  Other Names: SOS
  Arms: Soft occlusal splint group
Device: non-occlusive splint (NOS) — non-occlusive splint formed under vacuum from individual sheets of rigid polyethylene terephthalate 2 mm thick (Biolon, Dreve, Unna, Germany), from which the occlusal surfaces were cut and incisal edges, allowing the usual occlusal contact of each subject.
  Other Names: NOS
  Arms: Non-occlusive splint group

SUMMARY:
The objective of this study was to compare the clinical effectiveness of personalized thermoformed occlusal splints together with behavioral and self-care therapy in the management of myalgia of the masticatory muscles. A controlled clinical trial was carried out with a total of 46 subjects diagnosed with myalgia according to the diagnostic criteria for temporomandibular disorders (DC / TMD). All subjects were treated with behavioral and self-care therapy (BST) at the beginning of the study, and were then randomized into 4 groups: behavioral and self-care control group; rigid occlusal splint group; soft occlusal splint group and non-occlusive splint group. Follow-ups were carried out at 2, 6 and 10 weeks, where it was evaluated: pain in the masticatory muscles, mandibular range of motion, mandibular functional limitation and occlusal discomfort.

DETAILED DESCRIPTION:
Materials and method This randomized controlled clinical trial was conducted between October 2017 and January 2018 at the Dental Clinic of the Andrés Bello University (Viña del Mar, Chile). The study subjects were recruited from the universe of patients seeking treatment for jaw pain at the School of Dentistry. All subjects were informed about the study by their operator and gave their written consent before starting the study. The protocol, design and implementation were approved by the Scientific Ethics Committee of the Faculty of Dentistry of the Andrés Bello University, Viña del Mar, Chile (Folio No. 033, October 2017). Which was in accordance with the latest version of the Declaration of Helsinki of the World Medical Association (World Medical Association Declaration of Helsinki, 2013).

Sample Size Calculation It was calculated according to a confidence level of 95% and a statistical power of 80%. Based on a previous study by Niemelä et al. (Niemelä et al., 2012) it was determined that the variance of the main variable (masticatory muscle pain) of the reference group is 2.6. In turn, the pain variable was measured on the visual analog scale (VAS), where a minimum clinically relevant difference was considered if a 3.5 point decrease was achieved on the VAS scale with respect to treatment, a reference that was also considered in this study.

Randomization and interventions. After meeting the inclusion and exclusion criteria, the subjects were randomly assigned to four groups through a computationally generated sequence "list randomizer" developed by random.org.

Evaluation methods The initial evaluation, to determine the degree of involvement of axis I, was carried out following the symptom questionnaire and clinical examination guidelines according to the DC / TMD protocol. Additionally, the questionnaire for the chronic pain degree scale (GCPS v2.0) and the functional limitation scale (JFLS-20) of axis II of the DC / TMD protocol were applied. In turn, an intraoral clinical examination was performed to exclude pain of dental origin. No subject was excluded for odontogenic pain.

Statistic analysis The demographic characteristics of the sample were reported descriptively. The data studied were tested to determine normality by using the Shapiro-Wilk and Doornik-Hansen tests, data that were parametric, so they were analyzed with a mixed ANOVA test, a factorial part and a repeated means part for the variables degree of chronic pain, masticatory muscle pain, mandibular range of motion, functional limitation and occlusal discomfort. The level of significance used was established at p 0.05. All statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) version 17 software (IBM, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Presence of myalgia of the masticatory muscles with or without limitation of the mouth opening according to DC / TMD diagnostic criteria

Exclusion Criteria:

* Painful joint TMD
* History of treatment for TMD
* Recent history of facial or cervical trauma
* Current orthodontic treatment
* Tooth mobility secondary to periodontal disease
* Subjects with loss of more than two teeth other than third molars and / or premolars due to orthodontic indication
* Subjects with systemic musculoskeletal diseases or who are under analgesic treatment
* Subjects with a diagnosed intellectual disability who cannot express their will to participate in scientific research as established by law 20.584 of Chile

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Masticatory muscle pain initial evaluation | It was applied in the initial evaluation
  Pain intensity was measured using a visual analog scale. Subjects were asked to mark the intensity of pain perceived at the time of examination. This scale has a score from 0 to 10, with 10 being the greatest pain experienced by the patient
Masticatory muscle pain at 2 weeks | It was applied in week 2 of intervention.
  Pain intensity was measured using a visual analog scale. Subjects were asked to mark the intensity of pain perceived at the time of examination. This scale has a score from 0 to 10, with 10 being the greatest pain experienced by the patient
Masticatory muscle pain at 6 weeks | It was applied in week 6 of intervention.
  Pain intensity was measured using a visual analog scale. Subjects were asked to mark the intensity of pain perceived at the time of examination. This scale has a score from 0 to 10, with 10 being the greatest pain experienced by the patient
Masticatory muscle pain at 10 weeks | It was applied in week 10 of intervention.
  Pain intensity was measured using a visual analog scale. Subjects were asked to mark the intensity of pain perceived at the time of examination. This scale has a score from 0 to 10, with 10 being the greatest pain experienced by the patient

SECONDARY OUTCOMES:
Mandibular range of movement initial evaluation | It was applied in the initial evaluation
  Maximum opening of the mouth in an autonomous and comfortable way, that is, without feeling pain and not assisted by the operator, measured in millimeters from incisal edge to incisal edge in the anterior teeth, compensating for the overbite
Mandibular range of movement at 2 weeks | It was applied in week 2 of intervention.
  Maximum opening of the mouth in an autonomous and comfortable way, that is, without feeling pain and not assisted by the operator, measured in millimeters from incisal edge to incisal edge in the anterior teeth, compensating for the overbite
Mandibular range of movement at 6 weeks | It was applied in week 6 of intervention.
  Maximum opening of the mouth in an autonomous and comfortable way, that is, without feeling pain and not assisted by the operator, measured in millimeters from incisal edge to incisal edge in the anterior teeth, compensating for the overbite
Mandibular range of movement at 10 weeks | It was applied in week 10 of intervention.
  Maximum opening of the mouth in an autonomous and comfortable way, that is, without feeling pain and not assisted by the operator, measured in millimeters from incisal edge to incisal edge in the anterior teeth, compensating for the overbite
Mandibular functional limitation initial | It was applied in the initial evaluation
  Scale in charge of globally assessing masticatory limitation, vertical mobility limitation, verbal and non-verbal communication limitation, included within a 20-item instrument thanks to the survey of mandibular functional limitation of the DC / TMD. This scale has a score of 0 to 10, with 10 being a severe limitation
Mandibular functional limitation final | It was applied in week 10 of intervention.
  Scale in charge of globally assessing masticatory limitation, vertical mobility limitation, verbal and non-verbal communication limitation, included within a 20-item instrument thanks to the survey of mandibular functional limitation of the DC / TMD. This scale has a score of 0 to 10, with 10 being a severe limitation
Grade of chronic pain | It was applied in the initial evaluation
  The evaluation of the chronicity of the painful clinical picture and the disability that it involves was measured using the Graded Chronic Pain Scale of the DC / TMD, where I = Low intensity pain , without disability; II = High intensity pain, without disability; III = Moderate disability; IV = Severe disability.
Occlusal discomfort associated with an occlusal splint at 2 weeks | It was applied in week 2 of intervention.
  Scale responsible for evaluating adverse effects or discomfort of the subject to the occlusal splint during treatment, using a visual analog scale. This scale has a score of 0 to 10, with 10 being the greatest discomfort experienced by the patient.
Occlusal discomfort associated with an occlusal splint at 6 weeks | It was applied in week 6 of intervention.
  Scale responsible for evaluating adverse effects or discomfort of the subject to the occlusal splint during treatment, using a visual analog scale. This scale has a score of 0 to 10, with 10 being the greatest discomfort experienced by the patient.
Occlusal discomfort associated with an occlusal splint at 10 weeks | It was applied in week 10 of intervention.
  Scale responsible for evaluating adverse effects or discomfort of the subject to the occlusal splint during treatment, using a visual analog scale. This scale has a score of 0 to 10, with 10 being the greatest discomfort experienced by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Diego I De Nordenflycht, Principal Investigator — Universidad Nacional Andrés Bello
Locations (1):
- Universidad Nacional Andrés Bello, Viña del Mar, Chile

IPD SHARING:
Plan to Share IPD: Yes
All the collected individual participant data (IPD), study protocol, statistical analysis plan, informed consent form and a clinical study report will be shared, including results, discussion and bibliography studied.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One-year database availability period, starting on October 19, 2020
Access Criteria: Database will be shared in Open Security Foundation (OSF), a non-profit public organization founded as a support organization for open source security projects.
URL: https://osf.io/9xtmd/

REFERENCES:
- [Background] Niemela K, Korpela M, Raustia A, Ylostalo P, Sipila K. Efficacy of stabilisation splint treatment on temporomandibular disorders. J Oral Rehabil. 2012 Nov;39(11):799-804. doi: 10.1111/j.1365-2842.2012.02335.x. Epub 2012 Jul 19. PMID 22809314
- See also: The DC/TMD is intended for use in both clinical settings and applied research settings. — https://ubwp.buffalo.edu/rdc-tmdinternational/tmd-assessmentdiagnosis/dc-tmd/
- Available data/document: Study Protocol: 10.17605/OSF.IO/9XTMD — https://osf.io/9xtmd/ — Supporting information for this study is available in the open science framework (OSF): the data set of individual participants, study protocol, statistical analysis plan, and informed consent form.